CLINICAL TRIAL: NCT06788275
Title: Effect of Different Aerobic Exercise Methods in Cardiac Rehabilitation on Endothelial Function in Patients With Ischaemic Heart Disease and Study of the Associated Physiological Mechanisms (ENDO-R)
Brief Title: Aerobic Exercise-induced Effect on Endothelial Function in Patients With Ischaemic Heart Disease
Acronym: ENDO-R
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Sanitaria y Biomédica de Alicante (Network)
Collaborators: Universidad Miguel Hernandez de Elche (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI2023/154; ISABIAL (Registry Identifier: ISABIAL: 2023-0447 / CEIm: PI2023/154)
Record Dates: First submitted 2025-01-15; First posted 2025-01-23 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-01

CONDITIONS: Percutaneous Coronary Intervention (PCI); Acute Myocardial Infarction; Angina (Stable); Unstable Angina Pectoris; Cardiorespiratory Fitness; Ischaemic Heart Diseases
Keywords: Aerobic exercise; High-intensity interval training; Cardiac rehabilitation; Multicenter study; Coronary artery disease; Flow-mediated dilation; Nitroglycerin-mediated dilation; Mortality predictors
MeSH Terms: conditions — Angina, Stable; Angina, Unstable; Coronary Artery Disease | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: An external researcher will conduct central allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Moderate-intensity training (MIT) group (Experimental): Continuous exercise training on a cycle ergometer
  Interventions: Behavioral: Aerobic exercise (MIT)
- Short high-intensity interval training (HIIT) group (Experimental): High-intensity interval exercise performed on a cycle ergometer
  Interventions: Behavioral: Aerobic exercise (Short HIIT)
- Long high-intensity interval training (HIIT) group (Experimental): High-intensity interval exercise performed on a cycle ergometer
  Interventions: Behavioral: Aerobic exercise (Long HIIT)

INTERVENTIONS:
Behavioral: Aerobic exercise (MIT) — Patients allocated to the MIT group will train on a cycle ergometer three days a week for 12 weeks (36 sessions). They will cycle continuously between the first and second ventilatory thresholds. The duration of each exercise session will be set according to the estimated energy expenditure of the long HIIT and short HIIT groups for each training block (energy expenditure-adjusted exercise sessions). All sessions will be supervised, and patients will be asked to avoid additional exercise. They will be allowed to perform extra physical activity (e.g., light walking) according to medical recommendations.
  Other Names: MIT
  Arms: Moderate-intensity training (MIT) group
Behavioral: Aerobic exercise (Short HIIT) — Patients allocated to the Short HIIT group will train on a cycle ergometer three days a week for 12 weeks (36 sessions). They will perform from two to four 4-repetition sets of 1-min above the second ventilatory threshold. Patients will perform 1- and 3-min active recovery periods below the first ventilatory threshold between repetitions and sets, respectively. The total time spent at high intensity will range from eight to 16 min. All sessions will be supervised, and patients will be asked to avoid additional exercise training. They will be allowed to perform extra physical activity (e.g., light walking) according to medical recommendations.
  Other Names: Short HIIT
  Arms: Short high-intensity interval training (HIIT) group
Behavioral: Aerobic exercise (Long HIIT) — Patients allocated to the Long HIIT will train on a cycle ergometer three days a week for 12 weeks (36 sessions). They will perform from two to four 4-min high-intensity exercise bouts above the second ventilatory threshold separated by 4-min active recovery periods below the first ventilatory threshold. The total time spent at high intensity will range from eight to 16 min. All sessions will be supervised, and patients will be asked to avoid additional exercise training. They will be allowed to perform extra physical activity (e.g., light walking) according to medical recommendations.
  Arms: Long high-intensity interval training (HIIT) group

SUMMARY:
Endothelial dysfunction is one of the aetiological factors in ischaemic heart disease (IHD). Aerobic exercise is effective in improving endothelial function, as measured by flow-mediated dilation (FMD), in patients with IHD. Within the aerobic exercise methods, there is evidence showing that high-intensity interval training (HIIT) increases FMD to a greater extent than moderate-intensity training (MIT) in these patients. Notably, in a recent review, our research group found that only studies performing long bouts of HIIT (long HIIT: higher than 1 min) found a greater effect on FMD, while no differences were found in those studies using short bouts of HIIT (short HIIT: ≤ 1 min) and MIT. However, no experimental studies comparing the effect of long HIIT, short HIIT, and MIT on endothelial function, as well as other predictors of mortality, such as cardiorespiratory fitness, brain-derived neurotrophic factor (BDNF) levels or parasympathetic branch activity, have been performed. Therefore, the main objective of this project will be to compare the effect of the three aerobic exercise methods on endothelial function, as measured by FMD, in patients with IHD. Complementarily, the effect of aerobic exercise, depending on the exercise method, on different mortality predictors will be compared. For this purpose, a multicentre randomised study will be carried out (2 hospitals in Elche and one in Alicante). Assessors will be blinded to the patients allocation. Participants will be aware about their allocation in the experimental groups due to the nature of the study. A total of 132 men and women with IHD (66 per sex), diagnosed between three and 12 months before the start of the intervention, aged between 45 and 75 years, and without limitations for the practice of exercise training, will be recruited. All patients will train 3 days a week for 12 weeks. Participants will be assessed before the intervention (i.e., pre), at 6 weeks of training (i.e., mid) and after the intervention (i.e., post). Physiological and psychological variables will be registered in the assessment periods. Training intensity will be individually prescribed based on the cardiopulmonary exercise test (CPET). Intensity exercise will be adapted after the first part of the intervention. Analysis of covariance will be used to compare the values of the three groups after the intervention for the continuous variables, including the pre-intervention value as a covariate, while a logistic regression model will be used for the categorical variables.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 45 and 75 years.
* Diagnosed with acute myocardial infarction, unstable or stable angina.
* Treated with percutaneous coronary intervention, coronary artery bypass grafting, or conservative treatment.
* Event or intervention within 3 to 12 months prior to participation in the study.
* Fluency in speaking and reading Spanish.
* Residing in Elche or surrounding areas and able to attend evaluations and the exercise programme (not planning to be absent for more than one week during the programme).
* Functional Class I-II according to the New York Heart Association (NYHA) classification.
* No physical limitations for exercise.
* Stable optimal medical treatment.
* Physically inactive, defined as 1) not meeting the World Health Organization recommendations for both aerobic and strength exercise, and 2) not participating in a structured exercise programme at least 3 days per week for more than 3 months. Both conditions must be met for inclusion. Note: Casual walking is not considered grounds for exclusion.

Exclusion Criteria:

* Use of walking assistive devices.
* Treatment with chemotherapy for any type of cancer in the past 2 years.
* Hospitalisation in an intensive care unit in the past 6 months for reasons other than the ischaemic event.
* Acute myocardial infarction group IV Killip-Kimball.
* Obesity grade III (≥40.0 kg/m²).
* Medical contraindication for inclusion in an exercise programme.
* Diabetes with uncontrolled blood glucose levels.
* Poorly controlled hypertension: resting blood pressure > 180/110 mmHg.
* Chest pain with exertion or ST-segment changes suggestive of residual ischemia during ergometry. Residual ischemia.
* Severely reduced functional capacity on initial ergometry (<5 metabolic equivalent of task).
* Left ventricular ejection fraction less than 50%.
* Severe stenosis of the left main coronary artery (>50% significant disease).
* Severe aortic stenosis, left ventricular outflow tract obstruction (e.g., obstructive hypertrophic cardiomyopathy) or aortic dissection.
* Severe valvulopathy.
* Acute pulmonary embolism or deep vein thrombosis.
* Severe pulmonary hypertension.
* Acute heart failure.
* Acute endocarditis, myocarditis, or pericarditis.
* Acute or chronic renal insufficiency (estimated glomerular filtration rate <30 ml/min).
* Pulmonary fibrosis or interstitial disease (severe respiratory insufficiency or confirmed chronic obstructive pulmonary disease).
* Uncontrolled cardiac arrhythmias/hemodynamically unstable.
* Permanent or persistent/paroxysmal atrial fibrillation with episodes in the past 6 months.
* High-grade cardiac block.
* Presence of implantable devices: cardiac resynchronization therapy pacemaker, implantable cardioverter defibrillators, or pacemaker.
* Presence of ischaemic symptoms during the incremental exercise test performed before the intervention.
* Severe autonomic or peripheral neuropathy.
* Use of nitrates in pharmacological treatment.
* Any planned surgical or medical intervention during the study period.
* Plans to participate in or current participation in other studies that may interfere with this study.
* Current pregnancy or intention to become pregnant during the study period.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in endothelial function at 7 weeks | 7 weeks
  Endothelial function (i.e., endothelial-dependent dilation) will be assessed by brachial FMD.
Change from baseline in endothelial function at 14 weeks | 14 weeks
  Endothelial function (i.e., endothelial-dependent dilation) will be assessed by brachial FMD.
Change from baseline in endothelial-independent dilation at 7 weeks | 7 weeks
  Brachial NMD will be used to measure endothelial-independent dilation.
Change from baseline in endothelial-independent dilation at 14 weeks | 14 weeks
  Brachial NMD will be used to measure endothelial-independent dilation.
Change from baseline in peak cardiopulmonary parameters at 7 weeks | 7 weeks
  Participants will perform a symptom-limited CPET on a cycle ergometer.
Change from baseline in peak cardiopulmonary parameters at 14 weeks | 14 weeks
  Participants will perform a symptom-limited CPET on a cycle ergometer.
Change from baseline in aerobic efficiency at 7 weeks | 7 weeks
  Efficiency-related variables will be measured during the CPET.
Change from baseline in aerobic efficiency at 14 weeks | 14 weeks
  Efficiency-related variables will be measured during the CPET.
Change from baseline in resting serum BDNF concentration at 7 weeks | 7 weeks
  Blood samples will be obtained through an indwelling catheter placed in the antecubital vein before the CPET.
Change from baseline in resting serum BDNF concentration at 14 weeks | 14 weeks
  Blood samples will be obtained through an indwelling catheter placed in the antecubital vein before the CPET.
Change from baseline in exercise-induced effect on serum BDNF at 7 weeks | 7 weeks
  Blood samples will be obtained through an indwelling catheter placed in the antecubital vein before and after the CPET.
Change from baseline in exercise-induced effect on serum BDNF at 14 weeks | 14 weeks
  Blood samples will be obtained through an indwelling catheter placed in the antecubital vein before and after the CPET.

SECONDARY OUTCOMES:
Change from baseline in pulmonary function at 7 and 14 weeks | 7 and 14 weeks
  Pulmonary function will be measured by spirometry
Change from baseline in resting cardiopulmonary parameters at 7 and 14 weeks | 7 and 14 weeks
  Patients will be asked to rest for 5 min before stating the CPET.
Change from baseline in cardiopulmonary parameters at first and second ventilatory thresholds at 7 and 14 weeks | 7 and 14 weeks
  First and second ventilatory threshold during the CPET will be analysed blindly using the ventilatory equivalents method.
Change from baseline in cardiopulmonary variables measured during the recovery at 7 and 14 weeks. | 7 and 14 weeks
  Cardiopulmonary variables will be measured during the 3-min recovery period of the CPET.
Change from baseline in MacNew domains at 7 and 14 weeks | 7 and 14 weeks
  The MacNew heart disease health-related quality of life instrument will be used as a disease-specific quality of life questionnaire. The MacNew consists of 27 items that fall into three domains (a 13-item physical limitations domain scale, a 14-item emotional function domain scale, and a 13-item social function domain scale). Scoring of the MacNew is straightforward. The maximum possible score in any domain is 7 (high quality of life) and the minimum is 1 (poor quality of life).
Change from baseline in body composition at 7 and 14 weeks | 7 and 14 weeks
  Bioimpedance assessment will be conducted in fasting state.
Change from baseline in resting heart rate variability (HRV) at 7 and 14 weeks | 7 and 14 weeks
  HRV will be measured after an overnight fasting period at the same time of day
Change from baseline in ability to inhibit cognitive interference at 7 and 14 weeks | 7 and 14 weeks
  The Stroop test will be used to assess the ability to inhibit cognitive interference.
Change from baseline in echocardiographic variables at 7 and 14 weeks | 7 and 14 weeks
  A resting echocardiographic assessment will be performed before starting the CPET. The echocardiographic variables measured will be left ventricular end-diastolic diameter, septal and posterior wall thickness, left atrium dimension and volume, left ventricular ejection fraction (four-chamber and biplane Simpson's method, tricuspid annular plane systolic excursion, S' wave velocity, peak E and A wave velocities (in sinus rhythm), lateral and medial e' velocities, peak tricuspid regurgitation gradient, and velocity and gradient across the aortic valve.
Change from baseline in blood analysis variables at 14 weeks. | 14 weeks
  Blood samples will be obtained after at least a 10-hours period of fasting.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Centro de Investigación del deporte, Elche, Alicante
  - Instituto de Investigación Sanitaria y Biomédica de Alicante, Alicante

IPD SHARING:
Plan to Share IPD: Yes
The Instituto de Investigacion Sanitaria y Biomedica de Alicante (ISABIAL) Community in ZENODO. Depositing in ZENODO allows selecting the type of access for each file (open, embargoed; restricted; closed) and the license for use (Creative Commons Attribution 4.0 International, which requires citing the database and the original study, as well as mentioning any changes made; this is suggested at the institutional level for files identified with open access). It is important to note that the use of ZENODO is temporary, until it is viable to use the REPISALUD repository, from the Carlos III Health Institute, by the ISABIAL research community. At least two different files will be included: i) The one corresponding to the data set; ii) One or more files with complementary information about the characteristics of the variables and/or study metadata (project, authors, related publication, keywords, etc.).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: From November 2027 to November 2030

REFERENCES:
- [Background] Fuertes-Kenneally L, Blasco-Peris C, Casanova-Lizon A, Baladzhaeva S, Climent V, Sarabia JM, Manresa-Rocamora A. Effects of high-intensity interval training on vascular function in patients with cardiovascular disease: a systematic review and meta-analysis. Front Physiol. 2023 Jul 27;14:1196665. doi: 10.3389/fphys.2023.1196665. eCollection 2023. PMID 37576344